CLINICAL TRIAL: NCT03268083
Title: An Open-Label, Dose-Finding, Phase II Study to Evaluate the Immunogenicity and Safety of the Bioreactor-generated EV71 Vaccine in Pediatric Subjects Aged 3 to 6 Years and 2 to 35 Months Old
Brief Title: A Study to Evaluate the Immunogenicity and Safety of EV71 Vaccine in Pediatric Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enimmune Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EV-BR1501
Record Dates: First submitted 2016-08-04; First posted 2017-08-31 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Enterovirus Infections
Keywords: Foot-and-Mouth Disease; Vaccines; Hand, Foot and Mouth Disease; EV71 vaccine
MeSH Terms: conditions — Enterovirus Infections; Foot-and-Mouth Disease; Hand, Foot and Mouth Disease | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group A1 (Experimental): 3 to 6 years
  Interventions: Biological: EV71 vaccine ([0.5 μg total protein + adjuvant 150 μg AI(OH)3] per dose)
- Group A2 (Experimental): 3 to 6 years
  Interventions: Biological: EV71 vaccine ([1 μg total protein + adjuvant 150 μg AI(OH)3] per dose)
- Group A3 (Experimental): 3 to 6 years
  Interventions: Biological: EV71 vaccine ([1 μg total protein ] per dose)
- Group B1 (Experimental): 2 to 35 months
  Interventions: Biological: EV71 vaccine ([0.5 μg total protein + adjuvant 150 μg AI(OH)3] per dose)
- Group B2 (Experimental): 2 to 35 months
  Interventions: Biological: EV71 vaccine ([1 μg total protein + adjuvant 150 μg AI(OH)3] per dose)
- Group B3 (Experimental): 2 to 35 months
  Interventions: Biological: EV71 vaccine ([1 μg total protein ] per dose)

INTERVENTIONS:
Biological: EV71 vaccine ([0.5 μg total protein + adjuvant 150 μg AI(OH)3] per dose) — Two vaccinations at 28 days apart
  Arms: Group A1; Group B1
Biological: EV71 vaccine ([1 μg total protein + adjuvant 150 μg AI(OH)3] per dose) — Two vaccinations at 28 days apart
  Arms: Group A2; Group B2
Biological: EV71 vaccine ([1 μg total protein ] per dose) — Two vaccinations at 28 days apart
  Arms: Group A3; Group B3

SUMMARY:
The objectives of this study are to evaluate the immune response and safety profiles of two injections of EV71 vaccine administrated with or without adjuvant Al(OH)3 at 0.5-μg and 1-μg dose in children aged 3 to 6 years old and 2 to 35 months old infants/toddlers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children aged from 3 to 6 years old (i.e. ≥ 3 years old and < 7 years old) for Part A,and from 2 to 35 months old (i.e. ≥ 2 months old and < 36 months old) for Part B at the time of first vaccination.
2. Subject's guardians are able and willing to comply with study procedures and provide the signed informed consent.
3. Subject is able and can comply with the requirements of the protocol.
4. Subject with body temperature ≤38°C.

Exclusion Criteria:

1. Subject with previous known exposure to Enterovirus 71 (EV71).
2. Subject with a history of herpangina, hand-foot-mouth disease,and acute hemorrhagic conjunctivitis associated with enterovirus infection in the past 3 months.
3. Subject with gestation < 37 weeks.
4. Subject with birth weight <2.5 kg.
5. Subject with a history of hypersensitivity to vaccines, or a history of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
6. Family history of seizures or progressive neurological disease.
7. Family history of congenital or hereditary immunodeficiency.
8. Severe malnutrition or dysgenopathy.
9. Major congenital defects or serious chronic illness, including perinatal brain damage.
10. Subject diagnosed of having autoimmune disease (e.g., celiac disease, type I diabetes, lupus (SLE), juvenile dermatomyositis, scleroderma, juvenile idiopathic arthritis (JIA), immune (or idiopathic) thrombocytopenia purpura).
11. Bleeding disorder diagnosed by a doctor or significant bruising or hemostatic difficulties with IM injections or blood draws.
12. Any acute infections 7 days prior to administrating the first vaccination.
13. Use of any investigational product (including drug, vaccine) within 30 days prior to vaccination or planned use during the study period.
14. Administration of any vaccines within 14 days prior to randomization.
15. Use of immunoglobulins or any blood products within 3 months prior to vaccination or planned use during the study period.
16. Chronic administration (defined as > 14 days) of immunosuppressants or other immunomodulators or systemic corticosteroids within 6 months prior to vaccination or planned use during the study period.
17. Subjects who had ever received investigational EV-71 vaccine prior to randomization.
18. Under anti-tuberculosis prevention or therapy.
19. Any condition that in the opinion of the investigator may interfere with the evaluation of study objectives.

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Serum neutralizing antibody titers (NT) induced by the EV71 vaccine | Day 56
  Evaluate the immunogenicity change of serum neutralizing antibody titers induced by the EV71 vaccine from baseline on Day 56
Seroconversion rate (SCR) based on neutralizing antibody titers | Day 56
  Evaluate the immunogenicity change of SCR from baseline on Day 56
Serum neutralizing antibody titers (NT) induced by the EV71 vaccine | Day 28
  Evaluate the immunogenicity change of serum neutralizing antibody titers induced by the EV71 vaccine from baseline on Day 28
Serum neutralizing antibody titers (NT) induced by the EV71 vaccine | Day 196
  Evaluate the immunogenicity change of serum neutralizing antibody titers induced by the EV71 vaccine from baseline on Day 196
Seroconversion rate (SCR) based on neutralizing antibody titers | Day 28
  Evaluate the immunogenicity change of SCR from baseline on Day 28
Seroconversion rate (SCR) based on neutralizing antibody titers | Day 196
  Evaluate the immunogenicity change of SCR from baseline on Day 196

SECONDARY OUTCOMES:
Solicited adverse events | 7 days after each vaccination
Unsolicited adverse events | 28 days after each vaccination
The occurrence of overall adverse events (AEs) and serious adverse event (SAEs) | Day 0 to Day 196
The occurrence of EV 71 breakthrough infection after Visit 3 | Day 57 to Day 364
Serum neutralizing antibody titers (NT) induced by the EV71 vaccine | Day 364
  Evaluate the immunogenicity of serum neutralization antibody titer induced by the EV 71 vaccine on Day 364

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hung MC, Cho CY, Chen CJ, Lai CC, Wu KG. Immunogenicity and safety of an inactivated enterovirus A71 vaccine in children 3-6 years and 2-35 months of age- an open-label, randomized phase IIb clinical trial. Vaccine. 2019 Sep 3;37(37):5559-5566. doi: 10.1016/j.vaccine.2019.07.096. Epub 2019 Aug 6. PMID 31399275